CLINICAL TRIAL: NCT05646992
Title: OPRTUNTI: Offering Potential for Reproduction Through Transplantation of Uterus iN the Treatment of Infertility
Brief Title: Uterus Transplantation to Treat Infertility
Acronym: OPRTUNTI
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00166167
Record Dates: First submitted 2022-12-02; First posted 2022-12-12 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Uterine Factor Infertility
Keywords: Uterus/Transplantation; Uterus/Surgery; Vascularized Composite Allotransplantation (VCA); Immunosuppression; Mayer-Rokitansky-Küster-Hauser (MRKH); Allotransplantation; Humans; Female; Hysterectomy
MeSH Terms: interventions — Tacrolimus; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Uterus Transplant Recipient (Experimental): Uterus recipients, who are otherwise healthy, adult, genotypic females affected by uterine factor infertility, will undergo the surgically innovative uterus transplantation procedure combined with short-term use of conventional calcineurin inhibitor-based immunosuppression in to support a fetus to a viable delivery via Caesarian section.
  Interventions: Procedure: Uterine Allotransplantation; Drug: Tacrolimus; Drug: Imuran

INTERVENTIONS:
Procedure: Uterine Allotransplantation — Temporary allogenic uterus transplantation from a living donor with the goal of achieving pregnancy and delivering viable baby.
Drug: Tacrolimus — Used as daily immunosuppression. Started at 3mg twice daily (PO) on post-operative Day 1, adjusted to achieve serum trough concentrations of 8-10ng/ml.
  Other Names: FK506
Drug: Imuran — Used as daily immunosuppresion. 100 mg for total body weight less than 75 kg and 150 mg for total body weight greater than or equal to 75 mgs
  Other Names: Azathioprine

SUMMARY:
This research study will use uterus transplantation to treat uterine factor infertility, also known as the inability to bear children due to not having a uterus. The purpose of this study is to enable women seeking genetically-related children and the childbearing experience to experience pregnancy and birth a child. In this study, living donors will undergo surgery to give the donor's uterus to another woman. The woman who receives the transplant will take immunosuppression to keep the uterus and herself healthy. Because taking immunosuppressive medicine has side effects, uterus transplantation is intended to be temporary, lasting about 5 years.

The goals of the study are successful pregnancy and the birth of one, and possibly two, healthy babies per transplant patient. The uterus is to be removed and immunosuppression stopped following the birth of a child. Offspring are delivered by Caesarian section, at which time the transplant may also be removed.

Transplant candidates must have fertilized, frozen (cryopreserved) embryos at a Johns Hopkins facility before undergoing transplantation. Transplant candidates will be asked to identify candidates' potential uterus donor. Altruistic donors, or women who want to donate without knowing a potential recipient, may also participate. All potential donors will be screened to see if the donors are a good match for a recipient and are healthy enough to have the donation surgery.

Study Duration:

* Uterus Donors: Screening through about 12 months following the transplant operation.
* Uterus Recipients: Recipients may have the uterus for about 5 years. After the transplant is removed, the study team will ask for yearly follow-ups for another 5 years.
* Children born from transplanted uteruses: The study team asks to follow offspring yearly through age 21 years.

DETAILED DESCRIPTION:
This is a prospective clinical cohort study to establish temporary allogenic uterus transplantation as a feasible and effective reconstructive strategy for the treatment of uterine factor infertility.

Suitable candidates will proceed through as many as nine study stages:

* Stage 1: Telephone Screening Interview
* Stage 2: Blood Work Screening
* Stage 3: In Vitro Fertilization (IVF) & Embryo Cryopreservation
* Stage 4: Full Screening
* Stage 5: Transplantation
* Stage 6: Embryo Transfer
* Stage 7: Pregnancy to Childbirth
* Stage 8: Uterus Explantation
* Stage 9: Longitudinal Follow-Up

Potential participants will first be screened by phone for general eligibility, motivations for transplantation, and probable identification of a living donor. Potential donors will be interviewed by an Independent Living Donor Advocate to determine eligibility. Suitable candidates and candidates' potential living donors will then undergo blood work screening to determine if it's an acceptable pairing for donation and transplantation. Next, if the recipient does not already have embryos banked at a Johns Hopkins Hospital facility, she will participate in IVF and embryo cryopreservation per standard of care protocols. After a sufficient number of fertilized embryos have been successfully stored, the participant and her living donor will undergo full study screening. Donor/recipient pairs deemed suitable for transplantation based on screening results will be scheduled for and undergo transplant surgery. Post-uterus donation, the donor will be followed according to post-hysterectomy surgery patient care protocols. Post transplantation, the recipient will continue under the care of the study team as a transplant patient as well as under the care of gynecologists, obstetricians, and maternal fetal medicine experts. Depending on the transplant recipient's post-operative course, embryo transfer may be attempted as early as 2 months post-transplant. Should the patient become pregnant, obstetrics will follow the participant's and her fetus' progress. Whether or not the recipient successfully carries a pregnancy or births a child, uterus explantation is an anticipated endpoint of this protocol. Patients will be counseled that participants may have the transplant to birth up to two offspring or for about five years, whichever comes first, after which removal of the uterus should be considered.

Study data on uterus transplant recipients will be collected for 5 years post-transplantation under this protocol, or for the entire time the participant has the graft, plus five years post-explantation. All attempts will be made to collect data on the offspring born as a result of this protocol through the offspring's 21st birthday.

ELIGIBILITY:
INCLUSION CRITERIA -

Recipient Inclusion Criteria:

* Genotypic female of any race, color, or ethnicity.
* Uterine factor infertility.
* Aged 18-38 years at time of egg retrieval.
* Strong desire to undergo uterus transplant in order to become pregnant and give birth to a child.
* Embryo cryopreservation with embryos located at Johns Hopkins:

  * Has a minimum of 4-8 cryopreserved normal embryos following Preimplantation Genetic Screening (PGS-screening).

OR o Is willing to undergo egg retrieval, in vitro fertilization, and PGS-screening to cryopreserve a minimum of 4-8 normal embryos.

* Willingness to undergo embryo implantation after uterus transplantation to achieve pregnancy.
* In the opinion of the study team, makes a reasonable effort to identify and refer her own potential uterus donor to the study team.
* Completes the protocol informed consent form.
* Non-smoker, defined by having never smoked or having quit >6 consecutive months prior to screening.
* No co-existing medical condition which, in the opinion of the study team, could affect the immunosuppression protocol, surgical procedure, or ability to be pregnant or bear a child. (See Donor and Recipient Exclusion Criteria below. If the condition is amenable to treatment, the study team must agree that said condition should not significantly enhance the surgical risks of uterus transplantation.)
* Negative serum pregnancy test.
* Blood type compatible with donor.
* Negative crossmatch with donor.
* Patient agrees to comply with the protocol and states a dedication to the treatment regime.
* Agrees to uterus explanation following birth of a child and or 5 years without successful pregnancy.

Donor Inclusion Criteria:

* Genotypic female with an intact uterus.
* Medical history includes known successful pregnancy (e.g., gravid uterus).
* Aged 25 - 65 years.
* Consents to uterus donation and required pre-donation screening.
* For females of child-bearing potential: Negative serum pregnancy test.
* Blood type compatible with recipient.
* Negative crossmatch with recipient.

Donor and Recipient Inclusion Criteria:

* USA citizen or equivalent.
* No co-existing psycho-social problems (i.e., alcoholism, drug abuse).
* BMI ≤35

  o A higher BMI may be accepted at the discretion of the study team.
* Negative for HIV at transplant.
* Negative for malignancy for past 5 years.

EXCLUSION CRITERIA-

Donor and Recipient Exclusion Criteria:

* Positive for any of the following conditions:

  * Insulin-dependent diabetes mellitus.
  * Untreated sepsis.
  * HIV (active or seropositive).
  * Active tuberculosis.
  * Active Hepatitis B infection.
  * Active Hepatitis C infection.
  * Viral encephalitis.
  * Toxoplasmosis.
  * Current/recent (within 3 months of donation/screening consent) IV drug abuse.
  * Significant cardiac disease
  * Significant vascular disease o
* Sensitized recipients with high levels (50%) of panel-reactive Human Leukocyte Antigens (HLA) antibodies.
* Conditions that may impact the success of the surgical procedure or increase the risk of postoperative complications including inherited coagulopathies like Hemophilia, Von-Willebrand's disease, Protein C and S deficiency, Thrombocythemias, Thalassemias, Sickle Cell disease, etc.
* Mixed connective tissue diseases and collagen diseases that can result in poor wound healing after surgery.
* Severe neurologic deficits.
* Patients considered unsuitable per the consulted Psychiatric/Psychologic appraisal.
* A history of medical non-compliance.

Donor Only Exclusion Criteria:

* Previous injury to the uterus including giving birth by Cesarean section.
* History of radiation therapy to the abdominal area.
* Other medical conditions, as determined by the study physicians, that would preclude donation.

Recipient Only Exclusion Criteria:

• Conditions that, in the opinion of the study team, may expose the recipient to unacceptable risks under immunosuppressive treatment.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2033-02-28 (Estimated); Study Completion 2043-02-28 (Estimated)

PRIMARY OUTCOMES:
Successful delivery of viable baby | Uterus transplantation to 5 years post uterus transplantation
  Successful implantation of fertilized embryo which is then carried to term with the baby delivered by Cesarean section.

SECONDARY OUTCOMES:
Number of hazardous drinkers as assessed by Alcohol Use Disorders Identification Test-Concise (AUDIT-C) | Pre-Transplantation Screening through 5 years post uterus explantation
  A brief alcohol screen that reliably identifies patients who are hazardous drinkers or have active alcohol use disorders
Stress as assessed by the Brief Coping Orientation to Problems Experienced (COPE) | Pre-Transplantation Screening through 5 years post uterus explantation
  A 28 item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event.
Resilience as assessed by the Connor Davidson Resilience Scale (CD-RISC)-10 | Pre-Transplantation Screening through 5 years post uterus explantation
  A unidimensional self-reported scale consisting of 10-items measuring resilience.
Relationship quality as assessed by the Dyadic Adjustment Scale (DAS) [if having child with a partner] | Pre-Transplantation Screening through 5 years post uterus explantation
  A 32-item measure designed to assess the relationship quality of intact (married or cohabiting) couples.
Drug use as assessed by the Drug Abuse Screening Test (DAST) 10 Drug Use Questionnaire | Pre-Transplantation Screening through 5 years post uterus explantation
  A 10-item self-report instrument which assesses drug use, not including alcohol or tobacco use, in the past 12 months.
Depression as assessed by the Patient Health Questionnaire (PHQ-9) | Pre-Transplantation Screening through 5 years post uterus explantation
  A brief, self-administered questionnaire that assesses depression symptoms.
Overall health status as assessed by the Medical Outcome Study Short Form-36 (SF-36) | Pre-Transplantation Screening through 5 years post uterus explantation
  A 36 item survey used to assess overall health status using 8 scaled scores for Vitality, Physical functioning, Bodily pain, General health perceptions, Physical role functioning, Emotional role functioning, Social role functioning, and Mental health
PTSD as assessed by the Posttraumatic Stress Disorder Checklist (PCL-5 PTSD Checklist) | Pre-Transplantation Screening through 5 years post uterus explantation
  A 20-item self-report measure of the Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5) symptoms of Posttraumatic Stress Disorder PTSD
Anxiety as assessed by the General Anxiety Disorder (GAD)-7 | Pre-Transplantation Screening through 5 years post uterus explantation
  A 7-item self-report used to identify patients with anxiety.
Positive outcomes as assessed by the Post-Traumatic Growth Inventory (PTGI) | Pre-Transplantation Screening through 5 years post uterus explantation
  A 21-item self-report measure used to assess positive outcomes after extremely stressful and potentially traumatic events.
Life satisfaction as assessed by the Psychological Measures by Satisfaction with Life Scale (SWLS) | Pre-Transplantation Screening through 5 years post uterus explantation
  SWLS is a measure of life satisfaction. Uses scale to rate from 1-7, Where 1 indicates strongly disagree to 7 indicating strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Redett, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States